CLINICAL TRIAL: NCT00153946
Title: Multicenter Randomized Open-Label Comparison Study on the Efficacy and Safety of Argatroban Monotherapy With Argatroban-Edaravone Combination Therapy
Brief Title: Edaravone and Argatroban Stroke Therapy Study for Acute Ischemic Stroke
Acronym: EAST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Combination Therapy for Acute Ischemic Stroke Study Group (Other)
Collaborators: Japan Cardiovascular Research Foundation (Other)
Responsible Party: Takenori Yamaguchi, M.D., President Emeritus, National Cardiovascular Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EAST
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-05-14 (Estimated); Status verified 2008-05

CONDITIONS: Stroke
Keywords: Free Radical Scavenger; Selective Thrombin Inhibitor; Acute ischemic stroke (nonlacunar and noncardioembolic)
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Edaravone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): The patients who are allocated to Argatroban monotherapy
  Interventions: Drug: Edaravone
- B (Active Comparator): The patients who are allocated to Edaravone-Argatroban combination therapy
  Interventions: Drug: Edaravone

INTERVENTIONS:
Drug: Edaravone — 30mg/20mL vial, twice per day, not longer than two weeks

SUMMARY:
Edaravone, a free radical scavenger, is a novel neuroprotective agent, and argatroban is a selective thrombin inhibitor. Both the drugs were approved by the Japanese Government, and have frequently been used for the treatment of acute brain infarction in Japan. The effect of combination therapy of these drugs, however, has not yet been elucidated. This study will test the safety and efficacy of the combination therapy with these agents in patients with acute non-cardioembolic and non-lacunar ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke < 24 hours of onset
* Measurable neurological deficits caused by the present attack, ranging from 1 to 22 of NIHSS score on admission

Exclusion Criteria:

* Definite or possible cardiogenic brain infarction
* Definite lacunar infarction
* Prior ischemic stroke within 6 months
* Evidence of hemorrhagic brain infarction, epidural hematoma, intracerebral hematoma, or intraventricular hemorrhage
* Severe consciousness disturbances (semicoma to deep coma)
* Neurological signs clearing spontaneously
* Disability of 2 or more on mRS score before the index stroke aPTT being out of the normal range or 1.5 times longer than the pretreatment value
* If taking an oral anticoagulant, INR being 1.6 or more, or no INR data
* Treatment with urokinase, t-PA, heparin, ozagrel sodium, warfarin, or antiplatelet except for aspirin before enrollment
* Intravascular surgery, surgical operation, hyperbaric oxygen therapy, or hypothermia therapy before enrollment
* Serum creatinine >1.5 mg/dL
* Severe hepatic or cardiac disorders, infectious disorders, dehydration, etc.
* Neoplasm
* Pregnancy
* Hypersensitivity to test drugs

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 814 (Actual)
Dates: Start 2004-08; Primary Completion 2008-03 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale (MRS) score | at 3 months
Symptomatic intracranial hemorrhage | for the initial 3 weeks

SECONDARY OUTCOMES:
NIHSS score, JSS score, Barthel Index, modified Rankin Scale score | at various time-points
Various adverse effects | for the 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Takenori Yamaguchi, MD, PhD, Study Chair — National Cerebral and Cardiovascular Center, Japan; Takenori Yamaguchi, MD, PhD, Principal Investigator — National Cerebral and Cardiovascular Center, Japan
Locations (1):
- EAST Study Office c/o National Cardiovascular Center, Suita, Osaka, Japan

REFERENCES:
- [Background] Jin YJ, Mima T, Raicu V, Park KC, Shimizu K. Combined argatroban and edaravone caused additive neuroprotection against 15 min of forebrain ischemia in gerbils. Neurosci Res. 2002 May;43(1):75-9. doi: 10.1016/s0168-0102(02)00019-6. PMID 12074843
- [Derived] Kumagai N, Origasa H, Nagao T, Takekawa H, Okuhara Y, Yamaguchi T. Prognostic significance of smoking in patients with acute ischemic stroke within 3 months of onset. J Stroke Cerebrovasc Dis. 2013 Aug;22(6):792-8. doi: 10.1016/j.jstrokecerebrovasdis.2012.04.010. Epub 2012 May 24. PMID 22633681